CLINICAL TRIAL: NCT03485781
Title: Assessment of Hypoxic Brain Injury by Analyzing Propofol-induced EEG Changes
Brief Title: Propofol-induced EEG Changes in Hypoxic Brain Injury
Acronym: PROPEA3
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); Helsinki University Central Hospital (Other); Cerenion Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: 302/2016
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Cardiac Arrest
Keywords: EEG; Intensive Care; Propofol
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PROPEA3 is a prospective observational study investigating the recovery of propofol-induced EEG slow-wave activity and its association with neurological outcome after cardiac arrest.

DETAILED DESCRIPTION:
PROPEA3 is a prospective observational study investigating the recovery of propofol-induced EEG slow-wave activity and its association with neurological outcome after cardiac arrest. Comatose adult patients admitted to intensive care unit (ICU) after cardiac arrest are included. Patients with previous neurological disease expected to affect substantially EEG are excluded. The patients' relatives are asked for an informed written consent to participate. In the intensive care, the patients are sedated using continuous infusion of propofol while receiving temperature management/hypothermia treatment following the ICUs' common practice. EEG is recorded continuously from the admission to the ICU until 48 hours from the cardiac arrest. EEG slow-wave activity is determined offline by calculating the low-frequency (<1 Hz) power from the signal. The neurological recovery of the patients is defined 6 months after cardiac arrest from patient documents and/or by phone call to the patient/relative using Cerebral Performance Category. After the follow-up period patient or the relative is also asked to fill a survey (SF-36) to estimate the health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Comatose patients admitted to intensive care after cardiac arrest

Exclusion Criteria:

* Previous neurological disease expected to affect EEG substantially

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients admitted to intensive care in the study units.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
EEG slow-wave activity | 0-48 hours
  EEG slow-wave activity defined by the low-frequency (<1 Hz) signal power calculated continuously from the beginning of EEG measurement until 48 hours from cardiac arrest. The study investigates the association between the slow-wave activity and neurological outcome i.e. Cerebral Performance Category after 6 month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Kortelainen, MD, PhD, Principal Investigator — University of Oulu
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kortelainen J, Vayrynen E, Huuskonen U, Laurila J, Koskenkari J, Backman JT, Alahuhta S, Seppanen T, Ala-Kokko T. Pilot Study of Propofol-induced Slow Waves as a Pharmacologic Test for Brain Dysfunction after Brain Injury. Anesthesiology. 2017 Jan;126(1):94-103. doi: 10.1097/ALN.0000000000001385. PMID 27749312